CLINICAL TRIAL: NCT01528774
Title: Culture and Characterization of Circulating Tumor Cells (CTC) From Patients With Malignant Melanoma and Other Cancers
Brief Title: Culture and Characterization of Circulating Tumor Cells (CTC) in Melanoma and Other Cancers
Acronym: CTC
Status: Completed | Type: Observational
Sponsor: Wolfram Samlowski (Other)
Collaborators: TrueCells, LLC (Industry); Comprehensive Cancer Centers of Nevada (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Wolfram Samlowski, Physician, Comprehensive Cancer Centers of Nevada; Member, Developmental Therapeutics and Genitourinary Committee, US Oncology Research Clinical; Professor, University of Nevada, Reno, Comprehensive Cancer Centers of Nevada
Organization: Comprehensive Cancer Centers of Nevada (Other)
Other Study IDs: 12.01.015
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Melanoma
Keywords: Melanoma; Circulating Tumor Cells; Prostate cancer; Sarcoma; Renal Cancer; Pancreatic neuroendocrine cancer; Other solid tumor
MeSH Terms: conditions — Melanoma; Neoplastic Cells, Circulating; Prostatic Neoplasms; Sarcoma; Kidney Neoplasms; Somatostatinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood (up to 40 cc) collected in four 7.5 - 10 ml tubes. Serum samples may be stored frozen in a coded, de-identified format until DNA or RNA is extracted for assays to allow for batch processing. Samples will be consumed in the course of the research studies. Viable tumor cells may be grown as long-term cell lines.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Melanoma: Patients with histologically confirmed melanoma
  Interventions: Other: Blood Draw
- Prostate: Patients with histologically confirmed prostate cancer
  Interventions: Other: Blood Draw
- Solid tumors - other: Patients with histologically confirmed solid tumor cancers other than melanoma and prostate
  Interventions: Other: Blood Draw
- Benign Hematologic Conditions: Patients diagnosed with non-cancerous hematologic conditions
  Interventions: Other: Blood Draw
- Healthy Volunteers: Family members of patients undergoing treatment at Comprehensive Cancer Centers of Nevada, or other healthy volunteers
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Approximately 40 cc of blood will be drawn from participants at a time when they are having blood drawn for routine or treatment-related purposes. Sequential samples may be obtained in the same manner from selected patients to allow exploration of potential correlation of CTC with response to treatment, progression-free survival and overall survival.

SUMMARY:
The purpose of this study is to determine if circulating tumor cells (CTC) can be accurately detected and isolated from the blood of participants with melanoma using novel laboratory techniques. Blood samples will be collected from participants with melanoma, and also from participants with other solid tumor cancers and healthy volunteers for purposes of comparison.

Relevant information will be collected from participant's medical record and stored in a coded manner in a password-protected format. This information will be used to look for correlations of research results on blood samples to participant's medical condition. Test results will not be given to participants or their physicians. In some cases, CTC may be grown for long-term cell lines for further research.

DETAILED DESCRIPTION:
A strong correlation has been established between CTC and the progression of breast, colon and prostate cancers. The number of CTC appears to act as a prognostic marker for relapse and survival in a number of epithelial cancers. Unfortunately, current CTC assays are not effective in reliably detecting circulating melanoma cells and the assay procedures damage cells prohibiting further study.

This study is designed to evaluate the sensitivity and specificity of the TrueCells assay, a novel approach to isolate and preserve cells for further research.

Primary Objectives:

* Evaluate feasibility and reproducibility of isolation of CTC using TrueCells technology.
* Optimize quantitative CTC recovery
* Provide preliminary data concerning correlation of these measurements with other methods of CTC recovery such as immunofluorescence, lipid-based staining.

Secondary Objectives:

* Explore correlation of immunofluorescent CTC assay and TrueCells CTC cultures with response to treatment by objective and immune response criteria, progression free survival, 1 and 2-year survival landmarks, and overall survival in cancer patients.
* Attempt to isolate long-term tumor cell lines for evaluation of somatic gene mutations, and gene and protein expression patterns related to individual tumors (not intended to identify familial or inherited mutations), and to test drug and biologic sensitivity.
* Isolate plasma RNA and DNA to assess expression tumor-specific markers (e.g., tyrosinase, B-FRAF, V600E, etc.) and metastasis-associated genes (e.g., MSH-1, thymidylate synthase, etc.).
* Perform ongoing developmental testing to continue to develop and optimize novel technical approaches to facilitate isolation of intact CTC.

Methods:

Blood samples will be collected from patients with melanoma (200), prostate cancer (200), other solid tumor cancers (up to 400), benign hematologic conditions (100), and healthy volunteers (up to 100). Sequential samples will be obtained from selected patients during disease progression or treatment response to allow exploration of potential correlation of CTC with response to treatment, progression-free survival and overall survival. Samples will be immediately de-identified and assigned a numerical code, dated and sent to TrueCells, LLC. Once donated, sample ownership passes to TrueCells, LLC.

Research studies include:

* CTC independently counted using immunofluorescent staining of thick smear prepared from entire buffy coat of two tubes of blood (tubes 1 & 2), stained with appropriate primary pan-tumor monoclonal antibody or lipid markers with confirmatory secondary antibodies to exclude inadvertent inclusion of leukocyte and endothelial subsets and verify recognition of the patient's cancer.
* Leukocytes (containing CTC) isolated by density gradient centrifugation. The buffy coat is plated into TrueCells proprietary cell culture medium and tumor cells grown and propagated (tubes 3 & 4). Cell colonies enumerated and compared to number of colonies identified by immunofluorescent staining.
* In some cases CTC may be able to be grown as long-term cell lines. These cells may be subject to further analysis such as evaluation of somatic gene mutations as well as gene and protein expression patterns to identify characteristics of individual tumors as well as drug and biologic agent sensitivity. There may be additional future in vitro experimental applications for these de-identified early-passage cell lines that have not yet been identified or anticipated in this application.
* Plasma (byproduct of leukocyte isolation process from tubes 3 & 4) will be collected and temporarily frozen for DNA and RNA isolation for molecular assays of melanoma molecular markers and metastatic gene expression. These samples are consumed in the assay procedure.

Clinical information will be abstracted from medical records and de-identified and stored in a password-protected spreadsheet. Information to be collected includes age, gender, T, N, M status, other health conditions, serum LDH, any specific tumor markers (e.g. PSA), circulating tumor cells (if analyzed by commercial assay), somatic genetic mutations present in cancer (e.g. B-RAF V600E in melanoma patients) mitotic rate of tumor, date of tumor diagnosis, treatment history, date of regional and metastatic progression and date of death (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of melanoma, prostate cancer or other solid tumor malignancy; or benign hematologic disorder; or healthy volunteer.
* 18 years of age or older.
* Signed written informed consent.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients receiving treatment for cancer at Comprehensive Cancer Centers of Nevada. Healthy volunteers (family members of CCCN patients or other volunteers) will also be accepted for study control purposes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Circulating tumor cell (CTC) isolation and colony counts | 2 years

SECONDARY OUTCOMES:
Immunophenotyping, somatic (tumor-specific) DNA mutation analysis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Samlowski, MD, Principal Investigator — Comprehensive Cancer Centers of Nevada
Locations (1):
- Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada, United States